CLINICAL TRIAL: NCT06361758
Title: Second-line Treatment With CAdonilimab and LEnvatinib for Unresectable HCC: A Single Arm, Multicenter, Phase II Trial. (SCALE)
Brief Title: Second-line Treatment With CAdonilimab and LEnvatinib for Unresectable HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI has initiated a global multicenter Phase II clinical trial in the same direction, conducted by Akesobio.
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Sun Yat-sen University (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Hui-Chuan Sun, Director, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-326(2)
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: cadonilimab (anti PD-1/CTLA-4 bispecific antibody)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+Lenvatinib (Experimental)
  Interventions: Drug: Cadonilimab+Lenvatinib

INTERVENTIONS:
Drug: Cadonilimab+Lenvatinib — Cadonilimab (AK104): 15mg/kg Q3W iv D1 + Lenvatinib: 8 mg (body weight <60 kg) or 12mg (body weight ≥60 kg) orally QD. Eligible patients will receive AK104 plus Lenvatinib until disease progression or withdrawn ICF or death, whichever comes first.

SUMMARY:
This is an open-label, multi-center, single-arm, phase II study to evaluate the efficacy and safety of lenvatinib in combination with cadonilimab as second-line therapy in subjects with advanced hepatocellular carcinoma (HCC) who failed first-line standard therapy of immunotheray and antiangiogenic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent and be able to comply with the visit and related procedures required by the study protocol
* Age 18-75 years old, Male of Female
* ECOG PS 0-1
* histologically/cytologically or clinically (according to Chinese guidelines for primary liver cancer diagnosis and treatment (2022) criteria) confirmed initial diagnosis of HCC
* Not suitable for radical surgery and/or local treatment, BCLC stage C or stage B who failed local treatment
* Patients who progressed on first-line standard system therapy (Atezolizumab plus bevacizumab, sintilimab combined with bevacizumab, or Camrelizumab and Apatinib, only these three regimenes) or with intolerable toxicity ( except for immunotherapy intolerance)
* Child Pugh A-B7
* Expected survival time≥12 weeks
* At least one measurable lesion (RECIST 1.1)
* Enough organ and bone marrow function

Exclusion Criteria:

* Fibrolamellar sarcomatoid or mixed cholangiocarcinoma-hepatocellular carcinoma.
* Other anti-tumor therapies have been received after first-line systemic anti-tumor therapy.
* Have history of hepatic encephalopathy, or a history of liver transplantation.
* There are clinical symptoms requiring drainage of pleural fluid, ascites, pericardial effusion.
* People with acute or chronic active hepatitis B or hepatitis C, hepatitis B virus (HBV) DNA > 2000IU/ml or 10^4 copies /ml; Hepatitis C virus (HCV) RNA > 10^3 copies /ml; Hepatitis B surface antigen (HbsAg) and anti-HCV antibodies were both positive.
* Central nervous system metastasis.
* Previous bleeding from esophageal or fundus varices due to portal hypertension occurred within 6 months.
* Autoimmune immune disease.
* HIV infection.
* Pregnant women.
* The presence of any serious or uncontrolled systemic disease.
* Other acute or chronic diseases, psychiatric disorders or abnormal laboratory test values that may lead to the following results: increasing the risk associated with research or drug administration, or interfering with the interpretation of research results. The Investigator considers that there are other potential risks that are not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1 | Up to two years
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per mRECIST | Up to two years
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to mRECIST.
Disease control Rate (DCR) | Up to two years
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1 and mRECIST respectively.
Duration of response (DoR) | Up to two years
  Defined as the time from the first dose to disease progression or death in patients who achieve complete or partial response.
Progression-Free-Survival (PFS) | Up to two years
  Defined as the time between signing the informed consent form to the disease progression (according to RECIST v1.1 criteria) or death due to any cause.
Overall survival Overall survival (OS) | Up to three years
  Defined as the time between the first dose to death due to any causes.
Incidence of Adverse Events | Up to two years
  Adverse events (AEs) ; serious adverse events (SAEs); Treatment related Adverse events (TRAEs); Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Overall Officials: Huichuan Sun, Principal Investigator — Study Principal Investigator
Locations (3):
- China (3):
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Sun Yat-sen University Cancer Center), Guangzhou
  - Eastern Hepatobiliary Surgery Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No